CLINICAL TRIAL: NCT02311751
Title: Repetitive Transcranial Magnetic Stimulation (rTMS) for Executive Function Deficits in Autism Spectrum Disorder and Effects on Brain Structure: A Pilot Study
Brief Title: rTMS for Executive Function Deficits in Autism Spectrum Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Academic Health Science Centres (Other)
Responsible Party: Principal Investigator, Stephanie Ameis, Clinician Scientist, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 119/2013
Record Dates: First submitted 2014-11-25; First posted 2014-12-08 (Estimated); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism Spectrum Disorder; Executive Function; rTMS (Repetitive Transcranial Magnetic Stimulation); MRI (Magnetic Resonance Imaging); Healthy Subjects
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active rTMS (Active Comparator): Active treatment will be delivered at an intensity that is 90% of the resting motor threshold (RMT). Stimulation will be delivered at 20 Hz with 25 simulation trains of 30 stimuli each (i.e., 750 stimuli) and an intertrain interval of 30 sec. Treatment will be applied in sequential order bilaterally to the left and right dorsolateral prefrontal cortex (DLPFC). The order of bilateral stimulation (i.e. right then left or left than right) will be held constant for all 20 treatments.
  Intervention: Device: Repetitive Transcranial Magnetic Stimulation
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation
- Sham rTMS (Sham Comparator): Sham stimulation will be delivered using the same stimulation parameters and at the site of active treatment, but with only the side-edge resting on the scalp. The coil will be angled 45 degrees way from the skull in a single-wing tilt position. This method produces sound and some somatic sensation (e.g. contraction of scalp muscles) similar to those of active stimulation, but with minimal direct brain effects.
  Intervention: Device: Repetitive Transcranial Magnetic Stimulation
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation — rTMS is a non-invasive procedure involving the use of magnetic fields to stimulate nerve cells.
  Other Names: MagPro x100 series (Medtronic A/S, Copenhagen, Denmark)

SUMMARY:
In this study, the investigators will be examining the effects of repetitive transcranial magnetic stimulation (rTMS) on executive function deficits in individuals with autism spectrum disorder. Half of the participants will be chosen by chance to receive active rTMS stimulation while half will be chosen by chance to receive sham rTMS. Sham rTMS will feel the same as active rTMS only there will be no direct brain stimulation. This is necessary to ensure that active rTMS is efficacious in the enhancement of executive function in individuals with autism spectrum disorder. Based on results from a recently published pilot study, the investigators propose that active rTMS treatment will result in a significant improvement in working memory performance compared to sham rTMS treatment.

DETAILED DESCRIPTION:
This study is a randomized, double blind, sham controlled study to evaluate the efficacy of repetitive transcranial magnetic stimulation (rTMS) as a treatment for executive function deficits in individuals with autism spectrum disorder between 16 and 25 years of age. The study duration is approximately 3 months, with the rTMS sessions lasting for 4 weeks, 5 times a week, for about 1 hour each. Several scales will be used to assess for symptom severity and adaptive functioning. Cognition will be assessed using a validated battery.

This study also involves a type of brain imaging known as magnetic resonance imaging (MRI) at the beginning and at the end of the 4 weeks of daily rTMS to better understand the effects of rTMS on brain structure and function. Investigators will measure the size and connections of different parts of the brain to assess brain structure and blood flow while participants are completing some basic tasks to asses brain function.

ELIGIBILITY:
Inclusion Criteria Autism Spectrum Disorder (ASD):

* Are fluent in the English language
* Have a diagnosis of high functioning ASD (HF-ASD) (i.e., are verbal with an Intelligence Quotient (IQ) ≥ 70)
* Are competent to consent based on the subjects' ability to provide a spontaneous narrative description of the key elements of the study
* Are clinically stable as determined by their treating physician, with no medication changes over the past 4 weeks

Exclusion Criteria (ASD):

* Have a history of substance abuse or dependence in the last 6 months or have a positive urine toxicology screen
* Have a concomitant major medical or neurologic illness
* Have had a seizure in the past, or have a first-degree relative with epilepsy
* Have an abnormal clinical EEG
* Are pregnant or likely to get pregnant during the next 4 weeks
* Are clinically unstable
* Are on benzodiazepines or anticonvulsant medication
* Have a history of rTMS treatment.

Inclusion Criteria (Healthy Controls):

* Are fluent in the English language
* Competent to consent

Exclusion Criteria (Healthy Controls):

* Have a history of substance abuse or dependence in the last 6 months or have a positive urine toxicology screen
* Have a major medical or neurologic illness
* Have a diagnosed learning disorder or impaired academic or adaptive functioning on history
* Are pregnant
* Have an IQ < 80
* Have a psychiatric diagnosis on diagnostic interview assessments.

Ages: 16 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2018-05-04 (Actual); Study Completion 2018-05-04 (Actual)

PRIMARY OUTCOMES:
Change in accuracy on the Cambridge Neuropsychological Test Automated Battery (CANTAB) Spatial Working Memory Task | Baseline; Post rTMS (4 weeks after baseline); One month follow up ( 4 weeks after post rTMS); 6 month follow up (post rTMS); One year follow up (post rTMS)
  Specifically the investigators will evaluate the changes in spatial working memory scores before and after rTMS treatment.

SECONDARY OUTCOMES:
Change in scores on Behaviour Rating Inventory of Executive Functioning (A) (BRIEF) (A) | Baseline; Post rTMS (4 weeks after baseline); One month follow up ( 4 weeks after post rTMS); 6 month follow up (post rTMS); One year follow up (post rTMS)
  Specifically the investigators will evaluate the changes in executive function (EF) scores before and after rTMS treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie H Ameis, M.D., M.S.C, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addictions and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moxon-Emre I, Daskalakis ZJ, Blumberger DM, Croarkin PE, Lyon RE, Forde NJ, Tani H, Truong P, Lai MC, Desarkar P, Sailasuta N, Szatmari P, Ameis SH. Modulation of Dorsolateral Prefrontal Cortex Glutamate/Glutamine Levels Following Repetitive Transcranial Magnetic Stimulation in Young Adults With Autism. Front Neurosci. 2021 Oct 6;15:711542. doi: 10.3389/fnins.2021.711542. eCollection 2021. PMID 34690671
- [Derived] Ameis SH, Blumberger DM, Croarkin PE, Mabbott DJ, Lai MC, Desarkar P, Szatmari P, Daskalakis ZJ. Treatment of Executive Function Deficits in autism spectrum disorder with repetitive transcranial magnetic stimulation: A double-blind, sham-controlled, pilot trial. Brain Stimul. 2020 May-Jun;13(3):539-547. doi: 10.1016/j.brs.2020.01.007. Epub 2020 Jan 15. PMID 32289673
- See also: Information about research at the Centre for Addiction and Mental Health, Canada's largest mental health and addiction teaching — http://www.camh.net/research